CLINICAL TRIAL: NCT04977063
Title: Comparison of Gastrointestinal Transit Measurements for the Atmo Capsule With Those of the Gold Standard (SmartPill) in Gastroparesis and Slow Transit Constipation Patients
Brief Title: Atmo SmartPill Comparison in Gastroparetic and Slow Transit Constipation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atmo Biosciences Pty Ltd (Industry)
Collaborators: University of Western Sydney (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ETH01064
Record Dates: First submitted 2021-06-28; First posted 2021-07-26 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Gastroparesis; Slow Transit
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Intervention Model Description: Randomised control trial involving simultaneous ingestion of two medical devices - the Atmo gas capsule and SmartPill.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SmartPill and Atmo capsule (Other): The SmartPill and Atmo gas capsule will be tested simultaneously. This will allow the ability of the Atmo gas capsule to measure gastrointestinal transit time to be compared to the SmartPill. The order of swallowing will be randomised using a computer-generated list. The two capsules will be swallowed within 5 minutes of each other
  Interventions: Device: Atmo gas capsule; Device: SmartPill

INTERVENTIONS:
Device: Atmo gas capsule — The Atmo Gas Capsule measures the capsules location and motility/transit times through gas sensing capabilities
Device: SmartPill — The SmartPill measures the capsules location and motility/transit times through pH sensing

SUMMARY:
This study will compare gastrointestinal transit time measured by the SmartPill and the Atmo gas capsule in patients with gastrointestinal motility disorders. Both of these devices allow gastrointestinal transit time to be measured, however the SmartPill senses pH changes whereas the Atmo Capsule measures gas profiles. A total of 60 participants (30 diagnosed with gastroparesis, 30 with slow transit constipation) will attend Macarthur Clinical School at Western Sydney University after an overnight fast. Participants will consume a standardised meal before ingesting the SmartPill and Atmo Capsule. Each participant will carry a data receiver until passage of the capsules. Anatomical landmarks will be defined by pH changes (SmartPill) or oxygen profiles (Atmo Capsule). Statistical analysis will be performed via linear regression and degrees of agreement for measurements between the two devices. Primary end-points will be the agreement between gastric emptying, small intestinal and colonic transit times generated by the devices.

DETAILED DESCRIPTION:
The Atmo gas capsule is an ingestible, wireless, gas sensing capsule that is currently being developed and commercialised as a biomarker tool for gastrointestinal disorders. Following ingestion, the Atmo gas capsule transmits information about gases and temperature to an external receiver. The oxygen concentration profiles generated allow the passage of the capsule between aerobic (small intestine) and anaerobic (large intestine) to be characterised. The practical application of the Atmo Capsule is currently limited by the need to validate oxygen concentrations as a marker of position within the gastrointestinal tract. Preliminary studies using intestinal ultrasound have shown that migration of the Atmo capsule from the stomach to the duodenum, and its passage from terminal ileum to caecum, corresponds with major changes in oxygen concentration.

The SmartPill measures pH and offers gold-standard measurements of gastrointestinal transit times. To validate the ability of the Atmo Capsule to measure gastrointestinal transit time, this device will be compared to the SmartPill. This will allow the equivalence of these two devices in gastrointestinal transit measurements to be evaluated.

This study aims to compare gastrointestinal transit times using immediately sequential ingestion of the SmartPill and Atmo capsule in patients with gastrointestinal motility disorders. A total of 60 participants diagnosed with either gastroparesis (n=30) or slow transit constipation (n=30) will be recruited by advertisement (via online support group pages, such as Gastroparesis Australia) and word-of-mouth. Potential participants will be screened for eligibility. Suitable individuals will be sent a Participant Information Sheet and Consent Form for review. Participants will be asked to stop proton pump inhibitors, histamine receptor blockers and antacids 3 days prior to the study and during the study. Medications that affect gastric motility will also be stopped 48 hours before the start of the study and during the study. Following an overnight fast, participants will attend the Macarthur Clinical School, Western Sydney University, where the Principal Investigator (Dr Jerry Zhou) will review the Patient Information Sheet with each participant and obtain informed written consent. Participants will then be asked to consume a cereal bar with 200mL of water. Participants will subsequently ingest the SmartPill and Atmo capsule. The order of swallowing these devices will be randomised with a computer-generated list. Participants will be monitored for 15 minutes post-ingestion. Subjects will then fast for the next 6 hours, after which they will consume their normal meals for the rest of the day. The data receiver for both the SmartPill and Atmo capsule will be worn or kept within 1.5 metres of the body until passage of the capsule has been confirmed by observation in the toilet bowl or signal loss from both capsules after a bowel movement.

Adverse events, bowel movements and the presence of gastrointestinal symptoms will be recorded in a digital diary (as part of the Atmo receiver system) whilst the Atmo capsule is in the body. Once both devices have passed from the body, participants will attend Macarthur Clinical School, where receivers will be returned and an investigator will review the digital diary with them.The investigator will follow up with the participant via phone or email approximately one week after the study to enquire about symptoms and adverse effects.

For the SmartPill, anatomical landmarks will be identified by changes in pH profiles along the gastrointestinal tract as previously reported in the literature. More specifically, gastric emptying time will be defined by the time of capsule ingestion to the presence of a sharp rise in pH (more than three units), where the capsule passes from an acidic environment (pH ≤4) in the stomach to a more basic environment (pH >6) in the duodenum. Small intestinal transit will be determined by the time between the end of gastric emptying and identification of the ileo-caecal junction (a fall in ≥1 pH unit distal to gastric emptying). Colonic transit time will be defined as the time from ileocaecal junction to exit from the body. Whole gut transit time will be calculated as time of oral ingestion to exit from the body.

For the Atmo capsule, oxygen profiles will be used to characterise gastric emptying, small intestinal and colonic transit. Whole gut transit time will be calculated based on a change in temperature from exiting the body. The primary end-points of this study will be the agreement between gastric emptying, small intestinal and colonic transit times generated by the gas-sensing capsule vs wireless pH-motility. Statistical analysis with linear regression and by degrees of agreement (Bland-Altman tests) of measurements between the two devices will address these end-points. More subjects will be studied pending the results of this pilot study. The results, conduct and reporting of this study will conform to the STARD 2015 guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gastroparesis (idiopathic or diabetic) for at least 12 weeks (based on scintigraphy results) and able to eat orally.
* Diagnosed with slow transit constipation for at least 12 weeks (exclusion of constipation caused by structural abnormalities with colonoscopy, and confirmation of slow transit by 'marker studies' such as scintigraphy, radiolabelled or opaque X-ray study). Participant would have at least 1 bowel motion per week (either assisted or unassisted by medication).
* No evidence of metabolic disease (hypothyroidism, uncontrolled diabetes [hemoglobin A1c >10% within the past 6 months], electrolyte imbalance).
* An endoscopy or gastrointestinal barium series within the past 3 years showing no organic disease that is potentially causative of symptoms.
* Ability to stop medications that may alter gastric pH (such as proton pump inhibitors) for 3 days prior to and during study.
* Ability to stop medications that may alter gastrointestinal motility (GLP-1 angonists, anticholinergics, cannabinoids, metformin, antispasmodic, prokinetics) for 3 days prior to and during study.
* Ability to stop antibiotic, probiotic and, prebiotic supplements 7 days before prior to and during study.
* Ability to stop laxatives (docusate, lactulose, sorbitol, senna, bisacodyl), suppositories (glycerin), and enema 3 days prior to and during the study.
* Does not require a MRI scan during the duration of this study

Exclusion Criteria:

* Previous abdominal and/or pelvic surgery
* History of diverticulitis, diverticular stricture, and other intestinal strictures
* Chronic daily use of nonsteroidal anti-inflammatory drugs (ibuprofen, naproxen, etc.)
* Pregnant or nursing
* Patients on long-acting glucagon-like peptide (GLP-1)
* Implantable devices (e.g. pacemaker, defibrillator) [continuous glucose monitors are permitted].
* History of bezoar formation
* Dysphagia to solid foods
* Gastric/jejunal feeding tubes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Regional gastrointestinal metrics measured by Atmo gas capsule | 2 years
  Oxygen equivalence measured by the Atmo gas capsule will allow gastric emptying, small intestinal and colonic transit times to be determined.
Regional gastrointestinal metrics measured by SmartPill | 2 years
  pH data measured by the SmartPill will allow gastric emptying, small intestinal and colonic transit times to be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Zhou, PhD BSc, Principal Investigator — School of Medicine, Western Sydney University
Locations (3):
- Australia (3):
  - Blacktown Hospital, Blacktown, New South Wales
  - School of Medicine, Western Sydney University, Campbelltown, New South Wales
  - Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
Data will by only be available via manuscript for publication in an international peer reviewed journal.